CLINICAL TRIAL: NCT04136106
Title: The Incidence of Infection in Treatment of Low-dose IL-2 Combined With Corticosteroid and Immunosuppressor in SLE Patients- a Multi-center Prospective Study
Brief Title: The Incidence of Infection in Treatment of Low-dose IL-2 of SLE Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IL2Pro-01
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Infection
MeSH Terms: conditions — Infections | interventions — Interleukin-2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low-dose IL-2 group: Patients in this group were treated with low-dose IL-2 combined with corticosteroid and immunosuppressor, and low-dose IL-2 is defined as 100IU subcutaneously every other day for two weeks, followed by two-week break, as one treatment cycle, and at least three cycles.
  Interventions: Drug: IL-2
- Non IL-2 group: Patients in this group were only treated with corticosteroid and immunosuppressor,

INTERVENTIONS:
Drug: IL-2 — IL-2 is a medicine which can use in autoimmune disease, infection or cancer with different dose. Low-dose IL-2 preferentially used in autoimmune disease, such as SLE. Our enrolled SLE patients will divided into two groups depend on whether use IL-2 or not, combined with corticosteroid and immunosuppressor.
  Groups: Low-dose IL-2 group

SUMMARY:
IL-2 is a pleiotropic cytokine which can regulate or stimulate the differentiation and function of CD4+, CD8+ and NK cells. An opened-labelled trial and a retrospective study have indicated the incidence of infection is lower in the treatment of low-dose IL-2 combined with corticosteroid and immunosuppressor. We are going to conduct a multi-center prospective observational study to verify the above results.

DETAILED DESCRIPTION:
We are going to conduct a multi-center prospective observational study, and plan to enroll 500 SLE patients. Low-dose IL-2 is defined as 100IU IL-2 injected subcutaneously every other day for two weeks, followed by two-week break as one treatment cycle, and at least three weeks.There will be 250 patients in low-dose IL-2 group which treat with IL-2 combined with steroid and immunosuppressor. Non-IL-2 group is only treat with steroid and immunosuppressor. These patients are followed by every one month until get infected, otherwise, patients will be followed for two years. We focus on the type, positive microorganisms, grade and treatment of infection. Then, we will compare the differences of above parameters between these two groups.

ELIGIBILITY:
Inclusion Criteria:

* SLE patients diagnosed by the ACR Criteria of 1987;
* Treated with low-dose IL-2, corticosteroid and immunosuppressor for SLE.
* Consent to participate in this study.
* Regular follow-up for at least 2 years.

Exclusion Criteria:

* Other autoimmune disease;
* Without treatment of low-dose IL-2, corticosteroid and immunosuppressor for SLE.
* Mental disorder without regular or specific treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Depending on the incidence of infection in our retrospective study, Low-dose IL-2 group was 14.1%, non-IL-2 group was 25.2%. α was 0.05, β was 0.2, After the calculation of sample size, with the addition of about 20% patients for loss of follow-up, we plan to enroll 500 patients, and 250 patients in every groups equally.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of infection of two groups | 2 years
  Infection is confirmed by art least one infectious specialist or rheumatologist, by means of clinical symptoms, positive microorganisms culture, response to antibiotic therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, PhD,MD, Principal Investigator — Department of Rheumatology and Immunology, Peking University People's Hospital
Locations (1):
- Peking Universtiy People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] He J, Zhang X, Wei Y, Sun X, Chen Y, Deng J, Jin Y, Gan Y, Hu X, Jia R, Xu C, Hou Z, Leong YA, Zhu L, Feng J, An Y, Jia Y, Li C, Liu X, Ye H, Ren L, Li R, Yao H, Li Y, Chen S, Zhang X, Su Y, Guo J, Shen N, Morand EF, Yu D, Li Z. Low-dose interleukin-2 treatment selectively modulates CD4(+) T cell subsets in patients with systemic lupus erythematosus. Nat Med. 2016 Sep;22(9):991-3. doi: 10.1038/nm.4148. Epub 2016 Aug 8. PMID 27500725